CLINICAL TRIAL: NCT06613698
Title: A Dose-Finding, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of GSK4532990 for Steatohepatitis in Adults With Alcohol-related Liver Disease (ALD)
Brief Title: A Study to Investigate the Safety and Efficacy of GSK4532990 Compared With Placebo in Adult Participants Aged 18 to 65 Years With Alcohol-related Liver Disease
Acronym: STARLIGHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 222291; 2024-511596-15 (EudraCT Number)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Liver Diseases, Alcoholic
Keywords: GSK4532990; Alcohol-related liver disease; Steatohepatitis
MeSH Terms: conditions — Liver Diseases, Alcoholic; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- GSK4532990 Dose 1 (Experimental)
  Interventions: Drug: GSK4532990
- GSK4532990 Dose 2 (Experimental)
  Interventions: Drug: GSK4532990
- GSK4532990 Dose 3 (Experimental)
  Interventions: Drug: GSK4532990
- GSK4532990 Dose 4 (Experimental)
  Interventions: Drug: GSK4532990
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK4532990 — GSK4532990 will be administered
  Arms: GSK4532990 Dose 1; GSK4532990 Dose 2; GSK4532990 Dose 3; GSK4532990 Dose 4
Drug: Placebo — Placebo will be administered
  Arms: Placebo

SUMMARY:
The goal of this study is to assess the safety and efficacy of GSK4532990 in participants with alcohol-related liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent prior to the performance of any study-specific procedures.
* Able and willing to comply with all study assessments and adhere to the protocol schedule of activities.
* In the opinion of the investigator, there is a history of alcohol consumption compatible with either ALD or Met ALD.
* A female participant is eligible to participate after meeting additional pre-defined criteria.
* Participants must meet predefined stable use requirements of concomitant medications based on study criteria.

Exclusion Criteria:

* Meeting any definition of organ system failure as defined by the North American Consortium for Study of End-stage Liver Disease (NACSELD)
* Exceeding pre-defined biochemical parameters for Alanine Aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline Phosphatase (ALP), Platelets, International normalised ratio (INR), Albumin, estimated glomerular filtration rate (eGFR), Urine albumin-creatinine ratio (UACR) or Glycosylated Hemoglobin (HbA1c). Other primary causes of liver disease based on study criteria.
* Current malignancy (except for basal cell carcinoma or uterine carcinoma-in-situ) at screening. Participants under evaluation for possible malignancy at screening are not eligible.
* Prior organ transplant or current listing or active consideration for organ transplant during the screening period (except for corneal transplants).
* Chronic or acute, including partial, known portal vein thrombosis.
* Prior transjugular intrahepatic portosystemic shunt (TIPSS) insertion.
* Any acute cardiovascular event including myocardial infarction, unstable angina, symptomatic heart failure, or cerebrovascular accident in the 6 months prior to screening.
* Poorly controlled hypertension
* Clinical suspicion of rhabdomyolysis during the screening period
* Clinical suspicion of a bleeding episode during the screening period related to portal hypertension and/or low blood fibrinogen level.
* Body Mass Index (BMI) >35 kg/m2 at screening
* Any liver-related clinical event that started (onset) <8 weeks prior to Baseline (D1).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 8 weeks
Number of participants with potentially clinically relevant changes in electrocardiogram (ECG), vital signs, and clinical laboratory tests | Up to 8 weeks
Change from baseline in Liver Stiffness measurement (LSM) reduction using FibroScan® at Week 28 (kiloPascal) | Baseline (Day 1) and up to Week 28
  Liver stiffness will be measured by vibration-controlled transient elastography (VCTE) using the FibroScan® device.
Change from baseline in model for end-stage liver disease (MELD) score reduction at Week 28 | Baseline (Day 1) and up to Week 28
  MELD is a scoring system for assessing the severity of chronic liver disease. MELD scores range between 6 and 40, with 40 being the most severe.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of GSK4532990 | Up to Day 4
Area Under the Curve from Time 0 to t [AUC (0-t)] of GSK4532990 | Up to Day 4
Area Under the Curve from Time 0 to 24 hours [AUC (0-24)] of GSK4532990 | Up to 24 hours
Plasma half-life (t1/2) of GSK4532990 | Up to Day 4
Apparent clearance (CL/F) of GSK4532990 | Up to Day 4
Time to maximum concentration (tmax) of GSK4532990 | Up to Day 4
Apparent terminal phase volume of distribution (Vz/F) of GSK4532990 | Up to Day 4
Change from baseline in serum AST at Week 28 | Baseline (Day 1), and at Week28
Change from baseline in Enhanced Liver Fibrosis (ELF™) score at Week 28 | Baseline (Day 1), and at Week 28
  The ELF™ score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers, including tissue inhibitor of metalloproteinases-1 (TIMP-1), type III procollagen (PIIINP), and hyaluronic acid (HA). The ELF™ score is used as a prognostic marker for disease progression. ELF™ score will range between 4.5 to 14.7. A higher ELF™ score will predict worse prognosis
Area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC0-t) of GSK4532990 | Up to Day 3
Maximum observed plasma concentration (Cmax) of GSK4532990 | Up to Day 3

CONTACTS AND LOCATIONS:
Locations (101):
- United States (23):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Davis, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Parkville Melbourne, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Terrebonne, Quebec
- Denmark (3):
  - GSK Investigational Site, Esbjerg
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense C
- France (6):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Rouen
- Germany (4):
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Mainz
- Italy (6):
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Roma
- Japan (11):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (3):
  - GSK Investigational Site, DF
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
- GSK Investigational Site, Johannesburg, South Africa
- South Korea (5):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Gyeonggi-do
- Spain (8):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, León
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vigo
- Sweden (2):
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Kocaeli, İzmit
  - GSK Investigational Site, Diyarbakır, Sur
  - GSK Investigational Site, Adana, Yüreğir
  - GSK Investigational Site, Istanbul
- United Kingdom (8):
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Glasgow Strathclyde
  - GSK Investigational Site, Leeds West Yorkshire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/